CLINICAL TRIAL: NCT01356940
Title: A Randomized Controlled Double-blind Cross-over Trial of Dalfampridine ER for Effect on Ambulatory Activity in People With Multiple Sclerosis
Brief Title: A Placebo Controlled Trial of Dalfampridine ER for Ambulatory Activity in People With Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Principal Investigator, Theodore R Brown, Principle Investigator, Brown, Theodore R., M.D., MPH
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A randomized
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: Ambulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dalfampridine ER 10mg bid-placebo (Active Comparator): 4 week administration of dalfampridine ER 10mg bid followed by 2 week washout and 4 weeks of placebo control
  Interventions: Drug: dalfampridine ER; Drug: placebo
- placebo-dalfampridine ER 10mg bid (Placebo Comparator): placebo tablet administered bid for four weeks followed by 2 week washout and 4 weeks of dalfampridine ER 10mg bid
  Interventions: Drug: dalfampridine ER; Drug: placebo

INTERVENTIONS:
Drug: dalfampridine ER — dalfampridine ER 10mg bid for 4 weeks
  Other Names: Ampyra serial number 77948545
Drug: placebo — identical placebo tablet administered bid for four weeks
  Other Names: Sugar Pill

SUMMARY:
A randomized placebo controlled double-blind cross-over trial of Dalfampridine ER for effect on ambulatory activity in people with multiple sclerosis

DETAILED DESCRIPTION:
This is a parallel-group, double-blind, randomized controlled crossover trial with a 1:1 randomization. There are two treatment periods of 4 weeks and a two-week off treatment washout period. Treatment periods are DER (dalfampridine ER) followed by placebo (group A) and placebo followed by DER (group B), respectively. All dosages will be administered twice a week. Purpose of the study is to see if using the study drug(dalfampridine Er) for a short period of time will improve the way subjects with multiple sclerosis (MS) walk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS made at least 3 months prior to based McDonald or Proser criteria.
* Age 18-75 years old inclusive.
* Expanded Disability Status Scale (EDS) 0-6.5
* Clinical stability defined as no MS exacerbation or change in disease modifying therapy for 60 days prior to screening.
* Screening 6-minute walking test distance between 50m-500m, inclusive.
* Written informed consent.

Exclusion Criteria:

* use of 4-aminopyridine within 6 months of screening
* Any contraindication to DER:

  * Allergy to DER
  * history of seizure disorder or history of EEG showing epileptiform activity
  * Renal insufficiency (estimated GFR < 60.
* Any condition that would exclude 6 minute walking testing:

  * Cardiac surgery or myocardial infarction within the last 3 months.
  * Severe aortic stenosis or hypertropic cardiomyopathy.
  * Pulmonary embolus or infarction in the last 6 months.
  * Uncontrolled hypertension by history or by screening or baseline diastolic blood pressure > 170, or systolic blood pressure > 105.
  * Use of oxygen at home for 24 hours/day or severe lung disease.
* History of ventricular arrhythmia or finding of significant ventricular arrhythmia. atrial arrhythmia or 2nd or 3rd degree heart block on screening ECG.
* Concomitant neurological disease, such as ALS, Parkinson Disease, stroke.
* Hospitalization in the last 6 months for psychiatric illness.
* Alcohol or drug abuse within the past year.
* Females who are breast-feeding, pregnant or have potential to become pregnant during the course of the study( fertile and unwilling/unable to use effective contraceptive measures)
* Cognitive deficits that would interfere with the subject's ability to give informed consent or preform study testing.
* Any other serious and/or unstable medical condition.
* Use of mitoxantrone (Novantrone) within 6 months of baseline visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, Principal Investigator — EvergreenHealth
Locations (1):
- MS Center at Evergreen, Kirkland, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalfampridine ER 10mg Bid- Placebo: 4 week administration of dalfampridine ER 10mg bid followed by 2 week washout and 4 weeks of placebo
- Placebo-dalfampridine ER 10mg Bid: placebo tablet administered bid for four weeks followed by 2 week washout and dalfampridine ER: dalfampridine ER 10mg bid for 4 weeks
Period: First Intervention (28 Days)
Arm/Group | Dalfampridine ER 10mg Bid- Placebo | Placebo-dalfampridine ER 10mg Bid
Started | 22 | 21
Completed | 21 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout (14 Days)
Arm/Group | Dalfampridine ER 10mg Bid- Placebo | Placebo-dalfampridine ER 10mg Bid
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Second Intervention (28 Days)
Arm/Group | Dalfampridine ER 10mg Bid- Placebo | Placebo-dalfampridine ER 10mg Bid
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dalfampridine ER 10mg Bid Followed by Placebo: • Age 18-75 inclusive, Male or Female 4 week administration of dalfampridine ER 10mg bid
  Group A: dalfampridine ER 10mg bid for 4 weeks, 2 week washout, then matching placebo for 4 weeks
- Placebo Followed by Dalfampridine ER 10mg Bid: • Age 18-75 inclusive, Male or Female identical placebo tablet administered bid for four weeks
  Group B: identical placebo tablet administered bid for four weeks, 2 week washout, then dalfampridine ER 10mg bid for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Dalfampridine ER 10mg Bid Followed by Placebo | Placebo Followed by Dalfampridine ER 10mg Bid | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (2.5) | 53.3 (2.2) | 54.2 (2.3)
Sex/Gender, Customized [Number; unit: participants]
  female patients | 19 | 11 | 30
  male patients | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Peak Activity Index
Description: peak activity index is a measure of the 30 fastest minutes of walking over a 24 hour period, averaged over one week of accelerometer wear. Measurement is change from baseline to 4 weeks on intervention
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: change in strides per minute
Groups:
- Dalfampridine ER 10mg Bid: 4 week administration of dalfampridine ER 10mg bid
  dalfampridine ER: dalfampridine ER 10mg bid for 4 weeks
Arm/Group | Dalfampridine ER 10mg Bid | Placebo
Number analyzed (Participants) | 43 | 42
change in strides per minute | 0.6 (0.54) | 0.3 (0.55)
Statistical Analysis 1: Comparison: Dalfampridine ER 10mg Bid vs Placebo; Test type: Superiority or Other; p = 0.586, Mixed Models Analysis; Mean Difference (Final Values) = 0.586 — P values above 0.05 are considered statistically not significant in this study

2. Secondary Outcome: Stepcount
Description: change in daily stepcount recorded by an accelerometer and averaged over 1 week of wear baseline vs 4 weeks
Time Frame: 10 weeks
Population: total subject population
Measure: Least Squares Mean (Standard Deviation); unit: steps per day
Groups:
- Dalfampridine ER vs Baseline: 4 week administration of dalfampridine ER 10mg bid followed by 2 week washout and 4 weeks of placebo control
  dalfampridine ER: dalfampridine ER 10mg bid for 4 weeks
  placebo: identical placebo tablet administered bid for four weeks
- Placebo vs Baseline: placebo tablet administered bid for four weeks followed by 2 week washout and 4 weeks of dalfampridine ER 10mg bid
  dalfampridine ER: dalfampridine ER 10mg bid for 4 weeks
  placebo: identical placebo tablet administered bid for four weeks
Arm/Group | Dalfampridine ER vs Baseline | Placebo vs Baseline
Number analyzed (Participants) | 43 | 42
steps per day | 148.7 (222) | 128 (225)

ADVERSE EVENTS:
Arm/Group | Dalfampridine ER 10mg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 2/43 | 0/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalfampridine ER 10mg Bid (N=43) | Placebo (N=42)
worsening balance (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No